CLINICAL TRIAL: NCT02966522
Title: Frontline Thalidomide for Amyloidosis Involving Myocardium: Investigation of Organ Reversing Capacity of Lenalidomide
Brief Title: Thalidomide/Dexamethasone Treatment And PET Evaluation In Organ Involvemenet of Cardiac Amyloidosis
Acronym: TaPiOCA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: CW pharmaceutical company (Unknown)
Responsible Party: Principal Investigator, Youngil Koh, Clinical professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1512-129-730
Record Dates: First submitted 2016-11-08; First posted 2016-11-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cardiac Amyloidosis
Keywords: Thalidoide
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Thalidomide; Dexamethasone

ARMS (1):
- Thalidomide (Experimental): Patient with cardiac amyloidosis receive thalilomide with dexamethasone
  Interventions: Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Thalidomide
Drug: Dexamethasone

SUMMARY:
To prove the organ-reversing potential of thalidomide for amyloidosis with cardiac involvement

DETAILED DESCRIPTION:
Considering that dismal prognosis of amyloidosis is attributable to organ dysfunction, primary aim of amyloidosis treatment should be an organ reversal. However, due to various reasons, not much is known about organ reversal in amyloidosis. Almost all of the clinical trials evaluated hematologic response in amyloidosis. Meanwhile, besides autologous stem cell transplantation with high-dose melphalan conditioning, hematologic response rate of various agents such as bortezomib, melphalan, thalidomide and lenalidomide are similar for amyloidosis. However, organ reversing potential of these agents is not known. If there is a difference in organ reversing potential despite of similar hematologic response rate, drug with effective organ reversing potential should be a standard treatment for amyloidosis.

The investigators assume that thalidomide could make organ reversal in cardiac amyloidosis due to its specific mechanism of action. To prove this concept, the investigators propose a clinical trial that evaluates organ reversing potential of thalidomide in cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age : more than 18 years old
2. Cardiac amyloidosis (both AL or AH type) patient who meet both (A and B) of the following criteria A. Cardiac involvement: meet one of the following criteria

   * Echocardiography: mean wall thickness >12 mm, and no other cardiac cause
   * NTproBNP >332 ng/l in the absence of renal failure
   * Evidence of cardiac amyloidosis in cardiac MRI B. Treatment history: No history of exposure to thalidomide
3. ECOG(Eastern Cooperative Oncology Group) performance status ≤ 3
4. Tolerable major organ function determined by laboratory examination i. Serum creatinine ≤ 3.0 mg/dl ii. Absolute neutrophil count ≥ 1000/μl iii. Platelet ≥ 75000/ μl iv. Hemoglobin ≥ 8.0 mg/dl v. Bilirubin < 2 times or Alkaline phosphate < 4 times upper limit of normal
5. Expected survival > 3 months
6. Female participants of child-bearing potential must have a negative pregnancy test prior to treatment and agree to use dual methods of contraception for the duration of the study and for 30 days following completion of study. Male participants must also agree to use a barrier method of contraception for the duration of the study and for 30 days following completion of study if sexually active with a female of child-bearing potential.

Exclusion Criteria:

1. Amyloidosis without cardiac involvement
2. Patients who are planning to receive autologous stem cell transplantation
3. Patients who received autologous stem cell transplantation, remained in hematologic complete response
4. Pregnant, lactating or unwilling to use adequate contraception
5. Systemic infection unless specific anti-infective therapy is employed
6. Known allergies to thalidomide
7. Previous experimental agents or approved anti-tumor treatment within 1 months before the date of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Hematologic response | through study completion, an average of 1 year
  Complete response: Normalization of FLC levels and κ to λ ratio, with nega-tive serum and urine immunofixation Very good partial response: de-creased of dFLC to < 40mg/l Partial response: > 50% reduction of dFLC

SECONDARY OUTCOMES:
Cardiac response | through study completion, an average of 1 year
  > 30% and > 300 ng/l decrease in NTproBNP levels in patients with NTproBNP levels ≥ 650 ng/l at base-line or ≥ 2-class decrease in NYHA class in patients with NYHA class 3 or 4 at baseline
Maximal LV myocardium-blood cavity ratio | through study completion, an average of 1 year
  estimated by 11C-Pittsburge B PET imaging
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 60 months
Progression-free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Toxicity profile related to thalidomide, according to CTCAE version 4.03 | through study completion, an average of 1 year
Renal response | through study completion, an average of 1 year
  > 50% (≥ 5.0 g/d) decrease in 24h urine protein levels in patients with urine protein levels > 0.5 g/l at baseline without ≥ 25% increase in serum creatinine levels or decrease in creatinine clearance from baseline
Hepatic response | through study completion, an average of 1 year
  ≥ 50% decrease in alkaline phosphatase levels and/or ≥ 2cm decrease in liver size (assessed by radiograph)
Mean LV myocardium-blood cavity ratio | through study completion, an average of 1 year
  estimated by 11C-Pittsburge B PET imaging

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Kastritis E, Dimopoulos MA. Recent advances in the management of AL Amyloidosis. Br J Haematol. 2016 Jan;172(2):170-86. doi: 10.1111/bjh.13805. Epub 2015 Oct 22. PMID 26491974
- [Background] Gatt ME, Palladini G. Light chain amyloidosis 2012: a new era. Br J Haematol. 2013 Mar;160(5):582-98. doi: 10.1111/bjh.12191. Epub 2013 Jan 7. PMID 23294331
- [Background] Dispenzieri A, Buadi F, Laumann K, LaPlant B, Hayman SR, Kumar SK, Dingli D, Zeldenrust SR, Mikhael JR, Hall R, Rajkumar SV, Reeder C, Fonseca R, Bergsagel PL, Stewart AK, Roy V, Witzig TE, Lust JA, Russell SJ, Gertz MA, Lacy MQ. Activity of pomalidomide in patients with immunoglobulin light-chain amyloidosis. Blood. 2012 Jun 7;119(23):5397-404. doi: 10.1182/blood-2012-02-413161. Epub 2012 Apr 4. PMID 22493299
- [Background] Dispenzieri A, Lacy MQ, Zeldenrust SR, Hayman SR, Kumar SK, Geyer SM, Lust JA, Allred JB, Witzig TE, Rajkumar SV, Greipp PR, Russell SJ, Kabat B, Gertz MA. The activity of lenalidomide with or without dexamethasone in patients with primary systemic amyloidosis. Blood. 2007 Jan 15;109(2):465-70. doi: 10.1182/blood-2006-07-032987. Epub 2006 Sep 28. PMID 17008538
- [Background] Kastritis E, Terpos E, Roussou M, Gavriatopoulou M, Pamboukas C, Boletis I, Marinaki S, Apostolou T, Nikitas N, Gkortzolidis G, Michalis E, Delimpasi S, Dimopoulos MA. A phase 1/2 study of lenalidomide with low-dose oral cyclophosphamide and low-dose dexamethasone (RdC) in AL amyloidosis. Blood. 2012 Jun 7;119(23):5384-90. doi: 10.1182/blood-2011-12-396903. Epub 2012 Apr 18. PMID 22517904
- [Background] Lee SP, Lee ES, Choi H, Im HJ, Koh Y, Lee MH, Kwon JH, Paeng JC, Kim HK, Cheon GJ, Kim YJ, Kim I, Yoon SS, Seo JW, Sohn DW. 11C-Pittsburgh B PET imaging in cardiac amyloidosis. JACC Cardiovasc Imaging. 2015 Jan;8(1):50-59. doi: 10.1016/j.jcmg.2014.09.018. Epub 2014 Nov 4. PMID 25499132